CLINICAL TRIAL: NCT03629418
Title: Impact of Targeted Blood-pressure Management on Incidence of Acute Kidney Injury After Off-pump Coronary Artery Bypass Surgery: A Randomized Controlled Trial
Brief Title: Targeted Blood-pressure Management and Acute Kidney Injury After Coronary Artery Bypass Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anaesthesiology and Critical Care Medicine, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2018-118
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Coronary Artery Bypass, Off-Pump; Intraoperative Hypotension; Acute Kidney Injury; Preventive Medicine; Intraoperative Care
Keywords: Coronary Artery Bypass, Off-Pump; Intraoperative Hypotension; Acute Kidney Injury; Preventive Medicine; Intraoperative Care
MeSH Terms: conditions — Acute Kidney Injury | interventions — Norepinephrine; Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Targeted blood-pressure management (Experimental): Prophylactic norepinephrine infusion is started at the beginning of anesthetic induction and maintained throughout surgery. The target is to maintain systolic blood pressure at 110 mmHg or higher during surgery.
  Interventions: Drug: Targeted blood-pressure management
- Routine blood-pressure management (Active Comparator): Phenylephrine (25-50 ug) is injected or vasopressors is infused only when necessary. The target is to maintain systolic blood pressure at 90 mmHg or higher during surgery.
  Interventions: Drug: Routine blood-pressure management

INTERVENTIONS:
Drug: Targeted blood-pressure management — Prophylactic norepinephrine infusion is started before anesthetic induction and maintained throughout surgery. The target is to maintain systolic blood pressure at 110 mmHg or higher.
  Other Names: Norepinephrine
  Arms: Targeted blood-pressure management
Drug: Routine blood-pressure management — Phenylephrine (25-50 ug) is injected or vasopressors is infused only when necessary. The target is to maintain systolic blood pressure at 90 mmHg or higher during surgery.
  Other Names: Phenylephrine and other vasopressors
  Arms: Routine blood-pressure management

SUMMARY:
Acute renal injury (AKI) is a common complication after cardiac surgery and is associated with worse outcomes. It is now realized that intraoperative hypotension is an important risk factor for the development of AKI. In a recent randomized controlled trial of patients undergoing major noncardiac surgery, intraoperative individualized blood-pressure management reduced the incidence of postoperative organ dysfunction. The investigators hypothesize that, for patients undergoing off-pump CABG, targeted blood-pressure management during surgery may also reduce the incidence of postoperative AKI.

DETAILED DESCRIPTION:
Acute renal injury (AKI) is a common complication after cardiac surgery. In patients undergoing noncardiac surgery, intraoperative hypotension may lead to hypoperfusion of important organs and result in organ injuries such as AKI, myocardial injury, and stroke. The development of organ injuries is associated with wose outcomes including higher 30-day or even 1-year mortality. In a recent randomized controlled trial, patients undergoing major noncardiac surgery received either individualized (systolic blood pressure [SBP] maintained within 10% of the reference level) or standard (SBP maintained above 80 mmHg or within 40% of the reference level) blood-pressure management strategy during surgery. The results showed that individualized blood-pressure management reduced the incidence of postoperative organ dysfunction. Intraoperative hypotension is very common during off-pump coronary artery bypass grafting (CABG) surgery. The investigators hypothesize that, for patients undergoing off-pump CABG, good blood-pressure management with norepinephrine may also reduce the incidence of postoperative AKI. The purpose of this study is to investigate the effect of targeted blood-pressure management during off-pump CABG surgery on the incidence of postoperative AKI.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years;
* Scheduled to undergo off-pump CABG surgery.

Exclusion Criteria:

* Refuse to participate;
* Untreated or uncontrolled severe hypertension (systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥110 mmHg);
* Chronic kidney disease with a glomerular filtration rate < 30 ml/min/1.73 m2 or end-stage renal disease requiring renal-replacement therapy;
* Inability to communicate during the preoperative period because of coma, profound dementia, language barrier, or end-stage disease;
* Requirement of vasopressors/inotropics to maintain blood pressure before surgery;
* Second or emergency surgery;
* Expected survival of less than 24 hours.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 612 (Estimated)
Dates: Start 2018-08-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute kidney injury (AKI) within 7 days after surgery | Up to 7 days after surgery
  Development of AKI within 7 days after surgery is diagnosed according to the Kidney Disease Improving Global Outcomes (KDIGO) criteria

SECONDARY OUTCOMES:
Classification of AKI within 7 days after surgery | Up to 7 days after surgery
  Development of AKI within 7 days after surgery is diagnosed according to the KDIGO criteria
Incidence of delirium within 7 days after surgery | Up to 7 days after surgery
  Development of delirium within 7 days after surgery is assessed with the Confusion Assessment Method (3D-CAM for patients without mechanical ventilation and CAM-ICU for patients with mechanical ventilation).
Duration of mechanical ventilation after surgery | Up to 30 days after surgery
  Duration of mechanical ventilation after surgery
Length of stay in intensive care unit (ICU) after surgery | Up to 30 days after surgery
  Length of stay in intensive care unit (ICU) after surgery
Length of stay in hospital after surgery | Up to 30 days after surgery
  Length of stay in hospital after surgery
Incidence of major adverse cardiovascular events (MACEs) within 30 days after surgery | Up to 30 days after surgery
  MACEs within 30 days after surgery include cardiovascular death, non-fatal cardiac arrest, acute myocardial infarction, revascularization, and stroke.
Incidence of non-MACE complications within 30 days after surgery | Up to 30 days after surgery
  Non-MACE complications within 30 days after surgery indicate new-onset medical conditions other than MACEs that produce harmful effects on patients' recovery and required therapeutic intervention.
All-cause 30-day mortality | At 30 days after surgery
  All-cause 30-day mortality
2-year overall survival after surgery | Up to 2 years after surgery
  2-year overall survival after surgery
2-year major adverse cardiovascular event (MACE)-free survival after surgery | Up to 2 years after surgery
  MACEs within 2 years after surgery include cardiovascular death, non-fatal cardiac arrest, acute myocardial infarction, revascularization, and stroke.
Cognitive function in 1- and 2-year survivors | At the end of the 1st and 2nd years after surgery
  Cognitive function in 1- and 2-year survivors is assessed with the modified Telephone Interview for Cognitive Status (TICS-m, score ranges from 0 to 40, with higher score indicating better function).
Quality of life in 1- and 2- year survivors: SF-36 | At the end of the 1st and 2nd years after surgery
  Quality of life in 1- and 2-year survivors is assessed with the 36-Item Short Form Health Survey (SF-36). The SF-36 evaluates 8 different domains of quality of life, i.e., physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. The score of each domain ranges from 0 to 100, with high score indicating better function.

OTHER OUTCOMES:
Pain severity within 3 days after surgery: NRS | Up to 3 days after surgery
  Pain severity is assessed with the Numeric Rating Scale (NRS, an 11-point scale where 0=no pain and 10=the worst pain) twice daily (8:00-10:00 am, 18:00-20:00 pm) after surgery.
Daily prevalence of delirium during postoperative days 1-7 | During the first 7 days after surgery
  Daily prevalence of delirium during postoperative days 1-7
Duration of intraoperative cerebral desaturation (sub-study) | During surgery
  Duration of cerebral desaturation is monitored by near-infrared spectroscopy. Cerebral desaturation is defined as a decrease of more than 10% from baseline. Performed in part of enrolled patients.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Beijing University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abelha FJ, Botelho M, Fernandes V, Barros H. Determinants of postoperative acute kidney injury. Crit Care. 2009;13(3):R79. doi: 10.1186/cc7894. Epub 2009 May 22. PMID 19463152
- [Background] Bijker JB, van Klei WA, Vergouwe Y, Eleveld DJ, van Wolfswinkel L, Moons KG, Kalkman CJ. Intraoperative hypotension and 1-year mortality after noncardiac surgery. Anesthesiology. 2009 Dec;111(6):1217-26. doi: 10.1097/ALN.0b013e3181c14930. PMID 19934864
- [Background] Coca SG, Peixoto AJ, Garg AX, Krumholz HM, Parikh CR. The prognostic importance of a small acute decrement in kidney function in hospitalized patients: a systematic review and meta-analysis. Am J Kidney Dis. 2007 Nov;50(5):712-20. doi: 10.1053/j.ajkd.2007.07.018. PMID 17954284
- [Background] Monk TG, Saini V, Weldon BC, Sigl JC. Anesthetic management and one-year mortality after noncardiac surgery. Anesth Analg. 2005 Jan;100(1):4-10. doi: 10.1213/01.ANE.0000147519.82841.5E. PMID 15616043
- [Background] Schopka S, Diez C, Camboni D, Floerchinger B, Schmid C, Hilker M. Impact of cardiopulmonary bypass on acute kidney injury following coronary artery bypass grafting: a matched pair analysis. J Cardiothorac Surg. 2014 Jan 18;9:20. doi: 10.1186/1749-8090-9-20. PMID 24438155
- [Background] Rosner MH, Okusa MD. Acute kidney injury associated with cardiac surgery. Clin J Am Soc Nephrol. 2006 Jan;1(1):19-32. doi: 10.2215/CJN.00240605. Epub 2005 Oct 19. PMID 17699187
- [Background] Kheterpal S, Tremper KK, Heung M, Rosenberg AL, Englesbe M, Shanks AM, Campbell DA Jr. Development and validation of an acute kidney injury risk index for patients undergoing general surgery: results from a national data set. Anesthesiology. 2009 Mar;110(3):505-15. doi: 10.1097/ALN.0b013e3181979440. PMID 19212261
- [Background] Walsh M, Devereaux PJ, Garg AX, Kurz A, Turan A, Rodseth RN, Cywinski J, Thabane L, Sessler DI. Relationship between intraoperative mean arterial pressure and clinical outcomes after noncardiac surgery: toward an empirical definition of hypotension. Anesthesiology. 2013 Sep;119(3):507-15. doi: 10.1097/ALN.0b013e3182a10e26. PMID 23835589
- [Background] Bijker JB, Persoon S, Peelen LM, Moons KG, Kalkman CJ, Kappelle LJ, van Klei WA. Intraoperative hypotension and perioperative ischemic stroke after general surgery: a nested case-control study. Anesthesiology. 2012 Mar;116(3):658-64. doi: 10.1097/ALN.0b013e3182472320. PMID 22277949
- [Background] Rettig TCD, Peelen LM, Geuzebroek GSC, van Klei WA, Boer C, van der Veer JW, Hofland J, van de Garde EMW, Noordzij PG. Impact of Intraoperative Hypotension During Cardiopulmonary Bypass on Acute Kidney Injury After Coronary Artery Bypass Grafting. J Cardiothorac Vasc Anesth. 2017 Apr;31(2):522-528. doi: 10.1053/j.jvca.2016.07.040. Epub 2016 Jul 30. PMID 27727080
- [Background] Bennett-Guerrero E, Welsby I, Dunn TJ, Young LR, Wahl TA, Diers TL, Phillips-Bute BG, Newman MF, Mythen MG. The use of a postoperative morbidity survey to evaluate patients with prolonged hospitalization after routine, moderate-risk, elective surgery. Anesth Analg. 1999 Aug;89(2):514-9. doi: 10.1097/00000539-199908000-00050. PMID 10439777
- [Background] Hiltebrand LB, Koepfli E, Kimberger O, Sigurdsson GH, Brandt S. Hypotension during fluid-restricted abdominal surgery: effects of norepinephrine treatment on regional and microcirculatory blood flow in the intestinal tract. Anesthesiology. 2011 Mar;114(3):557-64. doi: 10.1097/ALN.0b013e31820bfc81. PMID 21307765
- [Background] Futier E, Lefrant JY, Guinot PG, Godet T, Lorne E, Cuvillon P, Bertran S, Leone M, Pastene B, Piriou V, Molliex S, Albanese J, Julia JM, Tavernier B, Imhoff E, Bazin JE, Constantin JM, Pereira B, Jaber S; INPRESS Study Group. Effect of Individualized vs Standard Blood Pressure Management Strategies on Postoperative Organ Dysfunction Among High-Risk Patients Undergoing Major Surgery: A Randomized Clinical Trial. JAMA. 2017 Oct 10;318(14):1346-1357. doi: 10.1001/jama.2017.14172. PMID 28973220
- [Background] Boettger S, Nunez DG, Meyer R, Richter A, Fernandez SF, Rudiger A, Schubert M, Jenewein J. Delirium in the intensive care setting and the Richmond Agitation and Sedation Scale (RASS): Drowsiness increases the risk and is subthreshold for delirium. J Psychosom Res. 2017 Dec;103:133-139. doi: 10.1016/j.jpsychores.2017.09.011. Epub 2017 Oct 4. PMID 29167040
- [Background] Chanques G, Garnier O, Carr J, Conseil M, de Jong A, Rowan CM, Ely EW, Jaber S. The CAM-ICU has now a French "official" version. The translation process of the 2014 updated Complete Training Manual of the Confusion Assessment Method for the Intensive Care Unit in French (CAM-ICU.fr). Anaesth Crit Care Pain Med. 2017 Oct;36(5):297-300. doi: 10.1016/j.accpm.2017.02.003. Epub 2017 Mar 29. PMID 28365244
- [Background] Katayama H, Kurokawa Y, Nakamura K, Ito H, Kanemitsu Y, Masuda N, Tsubosa Y, Satoh T, Yokomizo A, Fukuda H, Sasako M. Extended Clavien-Dindo classification of surgical complications: Japan Clinical Oncology Group postoperative complications criteria. Surg Today. 2016 Jun;46(6):668-85. doi: 10.1007/s00595-015-1236-x. Epub 2015 Aug 20. PMID 26289837